CLINICAL TRIAL: NCT01056965
Title: A 12 Week Randomized, Double Blind, Placebo-Controlled Pilot Study of Davunetide (NAP, AL-108) in Predicted Tauopathies
Brief Title: Davunetide (AL-108) in Predicted Tauopathies - Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Adam Boxer, Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL-108 NAP Pilot
Record Dates: First submitted 2010-01-21; First posted 2010-01-26 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Predicted Tauopathies, Including; Progressive Supranuclear Palsy; Frontotemporal Dementia With Parkinsonism Linked to Chromosome 17; Corticobasal Degeneration Syndrome; Progressive Nonfluent Aphasia
Keywords: Frontotemporal Dementia; Corticobasal Degeneration; Progressive Nonfluent Aphasia; Progressive Supranuclear Palsy; FTLD; FTD; PNFA; CBD; PSP; Predicted tauopathies, including:; Progressive Supranuclear Palsy (PSP); (CBS); Progressive Nonfluent Aphasia (PNFA)
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Primary Progressive Nonfluent Aphasia; Frontotemporal Dementia; Corticobasal Degeneration; Frontotemporal Lobar Degeneration | interventions — davunetide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- davunetide (Al-108, NAP) nasal spray (Experimental): Subjects will be randomized 2:1 (drug:placebo). Subjects will receive twice daily treatment with either davunetide 15 mg or placebo. Davunetide and placebo will be administered intranasally with a multi-dispensing, metered nasal spray pump device.
  Interventions: Drug: davunetide (AL-108, NAP)
- Placebo nasal spray (Placebo Comparator)
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: davunetide (AL-108, NAP) — Subjects will be randomized 2:1 (drug:placebo). Subjects will receive twice daily treatment with davunetide 15 mg administered intranasally.
  Other Names: AL-108; NAP
  Arms: davunetide (Al-108, NAP) nasal spray
Drug: Placebo nasal spray — Subjects will be randomized 2:1 (drug:placebo). Subjects will receive twice daily treatment with placebo administered intranasally.
  Arms: Placebo nasal spray

SUMMARY:
The primary objective of the study is to obtain preliminary safety and tolerability data with davunetide (NAP, AL-108) in patients with a tauopathy (frontotemporal lobar degeneration [FTLD] with predicted tau pathology, corticobasal degeneration syndrome [CBS] or progressive supranuclear palsy [PSP]). The secondary objectives of this study are to obtain preliminary data on short term changes (at 12 weeks) in a variety of clinical, functional and biomarker measurements from baseline, including cerebrospinal fluid (CSF) tau levels, eye movements, and brain MRI measurements.

ELIGIBILITY:
Inclusion Criteria:

1. A probable tauopathy defined as:

   * Probable or possible progressive supranuclear palsy (PSP) defined as:

     1. at least a 12-month history of:

        * postural instability or falls during the first 3 years that symptoms are present and
        * prominent decreased saccade velocity or supranuclear ophthalmoplegia;
     2. age at symptom onset ≥ 40 years by history; and
     3. an akinetic-rigid syndrome with prominent axial rigidity.

   OR,
   * Progressive nonfluent aphasia (PNFA)defined as:

     1. at least a 6-month history of difficulty with expressive speech characterized by at least 3 of the following:

        * apraxia of speech,
        * speech hesitancy,
        * labored speech,
        * word finding difficulty, or
        * agrammatism; and
     2. the symptoms above are the subject's principal neurological deficit and the symptoms constituted the initial clinical presentation.

   OR,
   * Corticobasal Degeneration syndrome (CBS) defined as:

     1. at least a 6-month history of progressive cortical dysfunction evidenced by at least one of the following:

        * ideomotor apraxia,
        * alien limb phenomenon,
        * cortical sensory loss,
        * focal or asymmetric myoclonus, or
        * apraxia of speech /nonfluent aphasia; and
     2. at least a 6-month history of progressive extrapyramidal dysfunction evidenced by at least one of the following:

        * focal or asymmetrical rigidity (limb or axial) or asymmetrical dystonia (limb or axial); and
        * lacking prominent and sustained L-dopa response.

   OR
   * Frontotemporal Dementia with Parkinsonism linked to Chromosome 17 (FTDP-17): Motor, cognitive or behavioral dysfunction, as defined below associated with a previously demonstrated mutation of the MAPT gene, and meets criteria for PNFA, CBS or PSP as defined above, or CDR-FTLD ≥ 1.0.
2. Documented age 40-85 years at the time of the onset of symptoms associated with the neurological deficits described in inclusion criterion 1.
3. Judged by investigator to be able to comply with neuropsychological evaluation at baseline.
4. Must have reliable caregiver accompany subject to all study visits. Caregiver must read, understand and speak local language fluently in order to ensure comprehension of informed consent form and informant-based assessments of subject. Caregiver must also have frequent contact with subject (at least 3 times per week for one hour) and be willing to monitor study medication compliance and the subject's health and concomitant medications throughout the study.
5. FTLD Modified Hachinski score ≤ 3.(Knopman et al., 2008) This modified Hachinski will not include the focal neurological signs, symptoms or pseudobulbar affect questions, given the prominence of all three in CBS/PSP.
6. MMSE ≥ 15 at Visit 1.
7. Written informed consent provided by both subject and caregiver who are both fluent English speakers.
8. Subject resides outside a skilled nursing facility or dementia care facility. Residence in an assisted living facility is allowed.
9. If the subject is receiving levodopa/carbidopa, a dopamine agonist, COMT inhibitor or other Parkinson's medication the dose must have been stable for at least 120 days prior to Visit 1 and must remain stable for the duration of the study.
10. Able to tolerate MRI scan during screening without use of sedation.
11. Able to ambulate with or without assistance.

Exclusion Criteria:

1. Insufficient fluency in local language to complete neuropsychological and functional assessments.
2. A diagnosis of Amyotrophic Lateral Sclerosis or other motor neuron disease.
3. Any of the following:

   * Abrupt onset of symptoms defined in inclusion criteria 1 associated with ictal events,
   * Head trauma related to onset of symptoms defined in inclusion criteria 1,
   * Severe amnesia within 6 months of the symptoms defined in inclusion criteria 1,
   * Cerebellar ataxia,
   * Choreoathetosis,
   * Early, symptomatic autonomic dysfunction, or
   * Tremor at rest.
4. History of other significant neurological or psychiatric disorders including, but not limited to, Alzheimer's disease, dementia with Lewy bodies, Prion disease, stroke, Parkinson's disease, any psychotic disorder, severe bipolar or unipolar depression, seizure disorder, tumor or other space-occupying lesion, or head injury with loss of consciousness within past 20 years temporally related to onset of symptoms.
5. Within 4 weeks of screening or during the course of the study, concurrent treatment with memantine (stable dose memantine, greater than 6 months is allowed), acetylcholinesterase inhibitors, antipsychotic agents or mood stabilizers (valproate, lithium, etc.) or benzodiazepines (other than temazepam or zolpidem).
6. Treatment with lithium, methylene blue, tramiprosate, ketone bodies, Dimebon or any putative disease-modifying agent directed at tau within 90 days of screening.
7. A history of alcohol or substance abuse within 1 year prior to screening and deemed to be clinically significant by the site investigator.
8. Any malignancy (other than non-metastatic basal cell carcinoma of the skin) within 5 years of Visit 1 or current clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal, or neurological disease. For the non-cancer conditions, if the condition has been stable for at least the past year and is judged by the site investigator not to interfere with the patient's participation in the study, the patient may be included.
9. Clinically significant lab abnormalities at screening, including creatinine ≥ 2.5 mg/dL, vitamin B12 below laboratory normal reference range, or TSH above laboratory normal reference range.
10. Systolic blood pressure greater than 180 or less than 90 mm Hg. Diastolic blood pressure greater than 105 or less than 50 mm Hg.
11. ECG abnormal at screening and judged to be clinically significant by the site investigator.
12. Treatment with any investigational drugs or device or participation in an investigational drug study within 60 days of screening.
13. Known history of serum or plasma progranulin level < 110.9 ng/mL.
14. Known presence of known disease-associated mutation in TDP-43, PGRN, CHMPB2 or VCP genes or any other FTLD causative genes not associated with underlying tau pathology (eg. Chr. 9 associated FTD).
15. History of deep brain stimulator surgery other than sham surgery for DBS clinical trial.
16. History of early, prominent REM behavior disorder.
17. Women of childbearing potential who are not using at least two forms of medically recognized contraception.
18. An employee or relative of an employee of Allon Therapeutics
19. Significant anatomical nasal abnormality (e.g., septal deviation obstructing airflow to at least one nostril or septal perforation) or history of nasal turbinate surgery.
20. History of a clinically significant medical condition that that would interfere with the subject's ability to comply with study instructions, would place the subject at increased risk, or might confound the interpretation of the study results.
21. Contraindication to MRI examination for any reason (eg., severe claustrophobia, ferromagnetic metal in body, etc.).
22. Structural abnormality on MRI within 2 years of baseline that precludes diagnosis of PSP, CBS or PNFA, such as cortical infarct in brain region that might account for subject's symptoms.
23. In subjects receiving anti-Parkinson's Disease medication at the time of screening, in the opinion of the investigator substantial worsening of motor signs or symptoms compared to normal functioning following overnight withdrawal of the anti-Parkinson medication.
24. Subject not willing to attempt LP.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety evaluations will be performed by recording clinical adverse events at each study visit. Clinical laboratory, ECGs, physical examinations will be conducted. | 12 weeks

SECONDARY OUTCOMES:
PSP Rating Scale | 12 weeks
Clinician's Global Impression (CGI-ds) | 12 weeks
Schwab and England Activities of Daily Living scale (SEADL) | 12 weeks
MRI brain ventricular volume | 12 weeks
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 12 weeks
Unified Parkinson's Disease Rating Scale (UPDRS) | 12 weeks
Neuropsychiatric Inventory (NPI) | 12 weeks
Geriatric Depression Scale (GDS) | 12 weeks
CSF biomarkers will assess total tau, phosphorylated tau, and amyloid beta peptide (1-42) | 12 weeks
Saccadic Eye movements - vertical and horizontal total saccade time | 12 weeks
Clinical Dementia Rating (CDR) | 12 weeeks
Functional Activities Questionnaire (FAQ) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adam L. Boxer, M.D., Ph.D., Principal Investigator — UCSF Memory and Aging Center
Locations (1):
- University of California, San Francisco (UCSF), San Francisco, California, United States

REFERENCES:
- [Background] Antoniades CA, Altham PM, Mason SL, Barker RA, Carpenter R. Saccadometry: a new tool for evaluating presymptomatic Huntington patients. Neuroreport. 2007 Jul 16;18(11):1133-6. doi: 10.1097/WNR.0b013e32821c560d. PMID 17589313
- [Background] Antoniades CA, Bak TH, Carpenter RH, Hodges JR, Barker RA. Diagnostic potential of saccadometry in progressive supranuclear palsy. Biomark Med. 2007 Dec;1(4):487-90. doi: 10.2217/17520363.1.4.487. PMID 20477368
- [Background] Bassan M, Zamostiano R, Davidson A, Pinhasov A, Giladi E, Perl O, Bassan H, Blat C, Gibney G, Glazner G, Brenneman DE, Gozes I. Complete sequence of a novel protein containing a femtomolar-activity-dependent neuroprotective peptide. J Neurochem. 1999 Mar;72(3):1283-93. doi: 10.1046/j.1471-4159.1999.0721283.x. PMID 10037502
- [Background] Bensimon G, Ludolph A, Agid Y, Vidailhet M, Payan C, Leigh PN; NNIPPS Study Group. Riluzole treatment, survival and diagnostic criteria in Parkinson plus disorders: the NNIPPS study. Brain. 2009 Jan;132(Pt 1):156-71. doi: 10.1093/brain/awn291. Epub 2008 Nov 23. PMID 19029129
- [Background] Boeve BF, Lang AE, Litvan I. Corticobasal degeneration and its relationship to progressive supranuclear palsy and frontotemporal dementia. Ann Neurol. 2003;54 Suppl 5:S15-9. doi: 10.1002/ana.10570. No abstract available. PMID 12833363
- [Background] Brenneman DE, Gozes I. A femtomolar-acting neuroprotective peptide. J Clin Invest. 1996 May 15;97(10):2299-307. doi: 10.1172/JCI118672. PMID 8636410
- [Background] Cairns NJ, Bigio EH, Mackenzie IR, Neumann M, Lee VM, Hatanpaa KJ, White CL 3rd, Schneider JA, Grinberg LT, Halliday G, Duyckaerts C, Lowe JS, Holm IE, Tolnay M, Okamoto K, Yokoo H, Murayama S, Woulfe J, Munoz DG, Dickson DW, Ince PG, Trojanowski JQ, Mann DM; Consortium for Frontotemporal Lobar Degeneration. Neuropathologic diagnostic and nosologic criteria for frontotemporal lobar degeneration: consensus of the Consortium for Frontotemporal Lobar Degeneration. Acta Neuropathol. 2007 Jul;114(1):5-22. doi: 10.1007/s00401-007-0237-2. Epub 2007 Jun 20. PMID 17579875
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Detre JA, Wang J, Wang Z, Rao H. Arterial spin-labeled perfusion MRI in basic and clinical neuroscience. Curr Opin Neurol. 2009 Aug;22(4):348-55. doi: 10.1097/WCO.0b013e32832d9505. PMID 19491678
- [Background] Dickson DW. Neuropathologic differentiation of progressive supranuclear palsy and corticobasal degeneration. J Neurol. 1999 Sep;246 Suppl 2:II6-15. doi: 10.1007/BF03161076. PMID 10525997
- [Background] Fahn S, Elton RL, Committee. Unified Parkinson's Disease Rating Scale. In: Fahn S, Marsden CD, Calne D and Goldstein M, editors. Recent Developments in Parkinson's Disease. Vol 2. Florham Park, NJ: Macmillan Health-care Information, 1987: 153-163.
- [Background] Furman S, Steingart RA, Mandel S, Hauser JM, Brenneman DE, Gozes I. Subcellular localization and secretion of activity-dependent neuroprotective protein in astrocytes. Neuron Glia Biol. 2004 Aug;1(3):193-9. doi: 10.1017/S1740925X05000013. PMID 16845437
- [Background] Garbutt S, Matlin A, Hellmuth J, Schenk AK, Johnson JK, Rosen H, Dean D, Kramer J, Neuhaus J, Miller BL, Lisberger SG, Boxer AL. Oculomotor function in frontotemporal lobar degeneration, related disorders and Alzheimer's disease. Brain. 2008 May;131(Pt 5):1268-81. doi: 10.1093/brain/awn047. Epub 2008 Mar 24. PMID 18362099
- [Background] Giladi E, Hill JM, Dresner E, Stack CM, Gozes I. Vasoactive intestinal peptide (VIP) regulates activity-dependent neuroprotective protein (ADNP) expression in vivo. J Mol Neurosci. 2007;33(3):278-83. doi: 10.1007/s12031-007-9003-0. Epub 2007 Oct 2. PMID 17952637
- [Background] Golbe LI, Ohman-Strickland PA. A clinical rating scale for progressive supranuclear palsy. Brain. 2007 Jun;130(Pt 6):1552-65. doi: 10.1093/brain/awm032. Epub 2007 Apr 2. PMID 17405767
- [Background] Gozes I, Brenneman DE. A new concept in the pharmacology of neuroprotection. J Mol Neurosci. 2000 Feb-Apr;14(1-2):61-8. doi: 10.1385/JMN:14:1-2:061. PMID 10854037
- [Background] Gozes I, Divinski I, Piltzer I. NAP and D-SAL: neuroprotection against the beta amyloid peptide (1-42). BMC Neurosci. 2008 Dec 10;9 Suppl 3(Suppl 3):S3. doi: 10.1186/1471-2202-9-S3-S3. PMID 19091000
- [Background] Gozes I, Divinsky I, Pilzer I, Fridkin M, Brenneman DE, Spier AD. From vasoactive intestinal peptide (VIP) through activity-dependent neuroprotective protein (ADNP) to NAP: a view of neuroprotection and cell division. J Mol Neurosci. 2003;20(3):315-22. doi: 10.1385/JMN:20:3:315. PMID 14501014
- [Background] Gozes I, Fridkinb M, Hill JM, Brenneman DE. Pharmaceutical VIP: prospects and problems. Curr Med Chem. 1999 Nov;6(11):1019-34. PMID 10519911
- [Background] Gozes I, Morimoto BH, Tiong J, Fox A, Sutherland K, Dangoor D, Holser-Cochav M, Vered K, Newton P, Aisen PS, Matsuoka Y, van Dyck CH, Thal L. NAP: research and development of a peptide derived from activity-dependent neuroprotective protein (ADNP). CNS Drug Rev. 2005 Winter;11(4):353-68. doi: 10.1111/j.1527-3458.2005.tb00053.x. PMID 16614735
- [Background] Kertesz A, Blair M, McMonagle P, Munoz DG. The diagnosis and course of frontotemporal dementia. Alzheimer Dis Assoc Disord. 2007 Apr-Jun;21(2):155-63. doi: 10.1097/WAD.0b013e31806547eb. PMID 17545742
- [Background] Knopman DS, Kramer JH, Boeve BF, Caselli RJ, Graff-Radford NR, Mendez MF, Miller BL, Mercaldo N. Development of methodology for conducting clinical trials in frontotemporal lobar degeneration. Brain. 2008 Nov;131(Pt 11):2957-68. doi: 10.1093/brain/awn234. Epub 2008 Oct 1. PMID 18829698
- [Background] Lee VM, Goedert M, Trojanowski JQ. Neurodegenerative tauopathies. Annu Rev Neurosci. 2001;24:1121-59. doi: 10.1146/annurev.neuro.24.1.1121. PMID 11520930
- [Background] Litvan I, Agid Y, Calne D, Campbell G, Dubois B, Duvoisin RC, Goetz CG, Golbe LI, Grafman J, Growdon JH, Hallett M, Jankovic J, Quinn NP, Tolosa E, Zee DS. Clinical research criteria for the diagnosis of progressive supranuclear palsy (Steele-Richardson-Olszewski syndrome): report of the NINDS-SPSP international workshop. Neurology. 1996 Jul;47(1):1-9. doi: 10.1212/wnl.47.1.1. PMID 8710059
- [Background] Mackenzie IR, Neumann M, Bigio EH, Cairns NJ, Alafuzoff I, Kril J, Kovacs GG, Ghetti B, Halliday G, Holm IE, Ince PG, Kamphorst W, Revesz T, Rozemuller AJ, Kumar-Singh S, Akiyama H, Baborie A, Spina S, Dickson DW, Trojanowski JQ, Mann DM. Nomenclature for neuropathologic subtypes of frontotemporal lobar degeneration: consensus recommendations. Acta Neuropathol. 2009 Jan;117(1):15-8. doi: 10.1007/s00401-008-0460-5. Epub 2008 Nov 18. No abstract available. PMID 19015862
- [Background] Matsuoka Y, Gray AJ, Hirata-Fukae C, Minami SS, Waterhouse EG, Mattson MP, LaFerla FM, Gozes I, Aisen PS. Intranasal NAP administration reduces accumulation of amyloid peptide and tau hyperphosphorylation in a transgenic mouse model of Alzheimer's disease at early pathological stage. J Mol Neurosci. 2007;31(2):165-70. doi: 10.1385/jmn/31:02:165. PMID 17478890
- [Background] Matsuoka Y, Jouroukhin Y, Gray AJ, Ma L, Hirata-Fukae C, Li HF, Feng L, Lecanu L, Walker BR, Planel E, Arancio O, Gozes I, Aisen PS. A neuronal microtubule-interacting agent, NAPVSIPQ, reduces tau pathology and enhances cognitive function in a mouse model of Alzheimer's disease. J Pharmacol Exp Ther. 2008 Apr;325(1):146-53. doi: 10.1124/jpet.107.130526. Epub 2008 Jan 16. PMID 18199809
- [Background] Neary D, Snowden JS, Gustafson L, Passant U, Stuss D, Black S, Freedman M, Kertesz A, Robert PH, Albert M, Boone K, Miller BL, Cummings J, Benson DF. Frontotemporal lobar degeneration: a consensus on clinical diagnostic criteria. Neurology. 1998 Dec;51(6):1546-54. doi: 10.1212/wnl.51.6.1546. PMID 9855500
- [Background] Oddo S, Caccamo A, Shepherd JD, Murphy MP, Golde TE, Kayed R, Metherate R, Mattson MP, Akbari Y, LaFerla FM. Triple-transgenic model of Alzheimer's disease with plaques and tangles: intracellular Abeta and synaptic dysfunction. Neuron. 2003 Jul 31;39(3):409-21. doi: 10.1016/s0896-6273(03)00434-3. PMID 12895417
- [Background] Pinhasov A, Mandel S, Torchinsky A, Giladi E, Pittel Z, Goldsweig AM, Servoss SJ, Brenneman DE, Gozes I. Activity-dependent neuroprotective protein: a novel gene essential for brain formation. Brain Res Dev Brain Res. 2003 Aug 12;144(1):83-90. doi: 10.1016/s0165-3806(03)00162-7. PMID 12888219
- [Background] Reed LA, Wszolek ZK, Hutton M. Phenotypic correlations in FTDP-17. Neurobiol Aging. 2001 Jan-Feb;22(1):89-107. doi: 10.1016/s0197-4580(00)00202-5. PMID 11164280
- [Background] Rivaud-Pechoux S, Vidailhet M, Gallouedec G, Litvan I, Gaymard B, Pierrot-Deseilligny C. Longitudinal ocular motor study in corticobasal degeneration and progressive supranuclear palsy. Neurology. 2000 Mar 14;54(5):1029-32. doi: 10.1212/wnl.54.5.1029. PMID 10720270
- [Background] Rosenmann H, Grigoriadis N, Eldar-Levy H, Avital A, Rozenstein L, Touloumi O, Behar L, Ben-Hur T, Avraham Y, Berry E, Segal M, Ginzburg I, Abramsky O. A novel transgenic mouse expressing double mutant tau driven by its natural promoter exhibits tauopathy characteristics. Exp Neurol. 2008 Jul;212(1):71-84. doi: 10.1016/j.expneurol.2008.03.007. Epub 2008 Mar 21. PMID 18490011
- [Background] Rottach KG, Riley DE, DiScenna AO, Zivotofsky AZ, Leigh RJ. Dynamic properties of horizontal and vertical eye movements in parkinsonian syndromes. Ann Neurol. 1996 Mar;39(3):368-77. doi: 10.1002/ana.410390314. PMID 8602756
- [Background] Schneider LS, Olin JT, Doody RS, Clark CM, Morris JC, Reisberg B, Schmitt FA, Grundman M, Thomas RG, Ferris SH. Validity and reliability of the Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S22-32. doi: 10.1097/00002093-199700112-00004. PMID 9236949
- [Background] Schwab R, England A. Projecton technique for evaluating surgery in Parkinson's disease. In: Gillingham F and Donaldson M, editors. Third Symposium on Parkinson's Disease Research. Edinburgh, Scotland: ES Livingston, 1969.
- [Background] Seeley WW, Crawford RK, Zhou J, Miller BL, Greicius MD. Neurodegenerative diseases target large-scale human brain networks. Neuron. 2009 Apr 16;62(1):42-52. doi: 10.1016/j.neuron.2009.03.024. PMID 19376066
- [Background] Shiryaev N, Jouroukhin Y, Giladi E, Polyzoidou E, Grigoriadis NC, Rosenmann H, Gozes I. NAP protects memory, increases soluble tau and reduces tau hyperphosphorylation in a tauopathy model. Neurobiol Dis. 2009 May;34(2):381-8. doi: 10.1016/j.nbd.2009.02.011. Epub 2009 Mar 2. PMID 19264130
- [Background] Smith-Swintosky VL, Gozes I, Brenneman DE, D'Andrea MR, Plata-Salaman CR. Activity-dependent neurotrophic factor-9 and NAP promote neurite outgrowth in rat hippocampal and cortical cultures. J Mol Neurosci. 2005;25(3):225-38. doi: 10.1385/JMN:25:3:225. PMID 15800376
- [Background] STEELE JC, RICHARDSON JC, OLSZEWSKI J. PROGRESSIVE SUPRANUCLEAR PALSY. A HETEROGENEOUS DEGENERATION INVOLVING THE BRAIN STEM, BASAL GANGLIA AND CEREBELLUM WITH VERTICAL GAZE AND PSEUDOBULBAR PALSY, NUCHAL DYSTONIA AND DEMENTIA. Arch Neurol. 1964 Apr;10:333-59. doi: 10.1001/archneur.1964.00460160003001. No abstract available. PMID 14107684
- [Background] Steingart RA, Solomon B, Brenneman DE, Fridkin M, Gozes I. VIP and peptides related to activity-dependent neurotrophic factor protect PC12 cells against oxidative stress. J Mol Neurosci. 2000 Dec;15(3):137-45. doi: 10.1385/JMN:15:3:137. PMID 11303778
- [Background] Vidailhet M, Rivaud S, Gouider-Khouja N, Pillon B, Bonnet AM, Gaymard B, Agid Y, Pierrot-Deseilligny C. Eye movements in parkinsonian syndromes. Ann Neurol. 1994 Apr;35(4):420-6. doi: 10.1002/ana.410350408. PMID 8154868
- [Background] Vulih-Shultzman I, Pinhasov A, Mandel S, Grigoriadis N, Touloumi O, Pittel Z, Gozes I. Activity-dependent neuroprotective protein snippet NAP reduces tau hyperphosphorylation and enhances learning in a novel transgenic mouse model. J Pharmacol Exp Ther. 2007 Nov;323(2):438-49. doi: 10.1124/jpet.107.129551. Epub 2007 Aug 24. PMID 17720885
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Zamostiano R, Pinhasov A, Gelber E, Steingart RA, Seroussi E, Giladi E, Bassan M, Wollman Y, Eyre HJ, Mulley JC, Brenneman DE, Gozes I. Cloning and characterization of the human activity-dependent neuroprotective protein. J Biol Chem. 2001 Jan 5;276(1):708-14. doi: 10.1074/jbc.M007416200. PMID 11013255
- [Background] Zusev M, Gozes I. Differential regulation of activity-dependent neuroprotective protein in rat astrocytes by VIP and PACAP. Regul Pept. 2004 Dec 15;123(1-3):33-41. doi: 10.1016/j.regpep.2004.05.021. PMID 15518891